CLINICAL TRIAL: NCT06879470
Title: An Early Exploratory Clinical Study on the Safety, Tolerability, and Preliminary Efficacy of JY231 Injection in the Treatment of Relapsed or Refractory B-Cell Lymphoma
Brief Title: JY231(JY231) Injection for the Treatment of Relapsed or Refractory B-Cell Lymphoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: He Huang (Other)
Responsible Party: Sponsor-Investigator, He Huang, Professor, Director of the Bone Marrow Transplantation Center, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JY-CT-24-006
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: B-Non Hodgkin Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A single-center, open, single arm study (Experimental): JY231 Injection for the treatment of relapsed or refractory B-cell lymphoma Subjects who meet the inclusion criteria will receive a single intravenous injection of JY231, followed by regular observation and follow-up of the subject.
  Interventions: Drug: JY231 Injection

INTERVENTIONS:
Drug: JY231 Injection — This is an open-label, single-arm study to evaluate the efficacy and safety of in vivo Chimeric Antigen Receptor T-Cell (CAR-T) therapy in patients with relapsed refractory B-cell leukemia.
  Upon enrollment, subjects will receive an intravenous infusion of the JY231 preparation. Following the infusion, subjects will be hospitalized for one month for observation, and subjects will be evaluated for safety and efficacy. Subjects will be followed for up to 15 years to determine if the disease is under control.

SUMMARY:
This study is an investigator-initiated single center, single arm clinical study with a target population of patients with relapsed or refractory B cell lymphoma. It is an early exploratory clinical study of the safety, tolerability and initial efficacy of JY231 injection in the treatment of relapsed or refractory B cell lymphoma.

DETAILED DESCRIPTION:
This study included the screening period (Day -18 to Day -7), the baseline period (Day -1), the treatment and observation period (Day 0 to 28), and the follow-up period (Month 2[from Day 29] to Year 15). Participants eligible for the screening period will be admitted to the study center for a single JY231 treatment and a follow-up period after the end of the treatment and observation period.

After completing the follow-up for the first five years, methods such as telephone or written questionnaires can be used, and relevant samples should be collected as much as possible. The subjects should be followed up at least once a year until the end of the follow-up period. The maximum monitoring time can be extended to 15 years, and all monitoring data during the extension process need to be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily signed an informed consent form and were willing and able to comply with all study requirements;
2. Age 18~75 years old, gender is not limited;
3. Malignant tumor cells positive for Cluster of Differentiation 19(CD19);
4. Meet the criteria for relapsed or refractory B-cell lymphoma. Relapsed: the subject's tumor reappears after achieving complete remission of the disease; refractory: the subject is ineffective or in only partial remission on standard treatment regimens. Subjects must have relapsed or become refractory after receiving at least two lines of systemic therapy or autologous hematopoietic stem cell transplantation.
5. The presence of at least one measurable lesion on imaging of relapsed or refractory B-cell lymphoma, i.e., a lymph node lesion >15 mm in length or an extranodal lesion >10 mm in length based on CT cross-sectional images, along with a positive Fluorodeoxyglucose Computed Tomography(FDG-PET).
6. Expected survival ≥12 weeks;
7. Eastern Cooperative Oncology Group(ECOG) score of 0 to 1 at baseline;
8. Good organ function (the standard can be appropriately relaxed for indicators involving liver and kidney function)

   1. Albuminous aminotransferase (ALT) ≤ 3 times the upper limit of normal (ULN);
   2. Albumin transaminase (AST) ≤ 3 times the ULN;
   3. Total bilirubin ≤ 1.5 times the ULN;
   4. Serum creatinine ≤1.5 times ULN or creatinine clearance ≥30 mL/min;
   5. Room oxygen saturation ≥92% without oxygen;
   6. left ventricular ejection fraction (LVEF) ≥50%;
9. Men of childbearing potential to ensure effective contraception for sexual partners; women of childbearing potential to use effective contraception and agree to use contraception throughout the study period.

Exclusion Criteria:

1. Subjects with active central nervous system (CNS) lymphoma;
2. Subjects with a history of active CNS disease such as seizures, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement;
3. Subjects who have been treated with another investigational drug within 30 days prior to screening or are still in the washout period;
4. Subjects who have had radiation therapy within 2 weeks prior to infusion;
5. Subjects with uncontrolled acute life-threatening bacterial, viral, or fungal infections (e.g., positive blood cultures ≤ 72 hours prior to infusion);
6. Subjects with unstable angina and/or myocardial infarction within 6 months prior to Screening;
7. Subjects with other prior or concurrent malignancies, with the following exceptions:

   1. Adequately treated basal cell, papillary thyroid, or squamous cell carcinoma (adequate wound healing is required prior to enrollment in the study);
   2. Carcinoma in situ of the cervix or breast, curatively treated, with no sign of recurrence for at least 3 years prior to study entry;
   3. Primary malignant tumor that has been completely resected and in complete remission for ≥ 5 years.
8. Presence of subjects with arrhythmias not controlled by medical management;
9. Subjects with active neurologic autoimmune or inflammatory conditions (e.g. Guillain-Barre syndrome, amyotrophic lateral sclerosis);
10. Women who are pregnant or breastfeeding, and female subjects who plan to become pregnant within 2 years of their JY231 injection infusion or male subjects whose partners plan to become pregnant within 2 years of their JY231 injection infusion;
11. Subjects who, in the investigator's judgment and/or clinical criteria, have a contraindication to any of the study procedures or have other medical conditions that may place them at unacceptable risk.
12. Other conditions that, in the opinion of the investigator, should not be enrolled in this clinical study, such as poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events(AE) after infusion | Day 28、Month 2、Month 3、Month 6、Month 12、Month 18、Month 24
  The frequency, severity, and laboratory findings of all adverse events/serious adverse events are included.
Maximal Tolerated Dose(MTD) | Up to 28 days after infusion
  MTD will be determined based on Dose-Limiting Toxicity(DLTs) observed during the first 28 days of study treatment.

SECONDARY OUTCOMES:
Objective Response Rate | Day 28、Month 2、Month 3、Month 6、Month 12、Month 18、Month 24
  Objective Response Rate(ORR) is defined as the proportion of subjects achieving complete remission(CR) and partial response(PR)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No